CLINICAL TRIAL: NCT02207569
Title: Medtronic CoreValve Evolut R United States IDE Clinical Study
Brief Title: Medtronic CoreValve Evolut R U.S. Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10126779DOC
Record Dates: First submitted 2014-07-24; First posted 2014-08-04 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CoreValve Evolut R TAVR system (Experimental): The CoreValve Evolut R System is a transcatheter aortic valve implantation system comprised of the following three components:
  1. Evolut R Transcatheter Aortic Valve (TAV)
  2. EnVeo R Delivery Catheter System (DCS) with EnVeo R InLine Sheath
  3. EnVeo R Loading System (LS)
  Interventions: Device: CoreValve Evolut R TAVR system

INTERVENTIONS:
Device: CoreValve Evolut R TAVR system

SUMMARY:
The study objectives are to assess the safety and efficacy of the CoreValve Evolut R transcatheter aortic valve replacement (TAVR) system in patients with severe symptomatic aortic stenosis are considered at high or extreme risk for surgical aortic valve replacement.

DETAILED DESCRIPTION:
This objective will be accomplished by a prospective, single arm, historical controlled, multi-site study involving a minimum of 150 implanted subjects with no more than 250 implanted subjects at up to 25 study sites in the United States. Procedural and 30 day safety and efficacy results from this study will be compared to appropriate historical control data for the Medtronic CoreValve System. Subjects will be followed up to 5 years following implantation.

The enrollment phase of the study is estimated to take approximately 6-9 months. As each implanted subject is to be followed up to 5 years, the estimated study duration is approximately 66-69 months, excluding the time required for preparing the final report.

ELIGIBILITY:
Inclusion Criteria - Severe aortic stenosis, defined as aortic valve area of < 1.0 cm2 (or aortic valve area index of < 0.6 cm2/m2) by the continuity equation, AND mean gradient > 40 mmHg or maximal aortic valve velocity > 4.0 m/sec by resting echocardiogram.

Subjects with low-flow/low gradient severe aortic stenosis can be included, provided low-dose dobutamine or exercise stress echocardiography demonstrates a mean gradient of >40 mmHg or a maximal aortic valve velocity of >4.0 m/sec, AND aortic valve area of <1.0cm2 (or aortic valve area index of <0.6 cm2/m2).

* STS score of ≥ 8 OR documented heart team agreement of ≥ high risk for AVR due to frailty or co-morbidities.
* Symptoms of aortic stenosis, AND NYHA Functional Class II or greater
* The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Exclusion Criteria

* Any condition considered a contraindication for placement of a bioprosthetic valve (e.g. subject is indicated for mechanical prosthetic valve).
* A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: aspirin or heparin (HIT/HITTS) and bivalirudin, ticlopidine and clopidogrel, Nitinol (titanium or nickel), contrast media
* Blood dyscrasias as defined: leukopenia (WBC < 1000 mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states.
* Untreated clinically significant coronary artery disease requiring revascularization.
* Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20% by echocardiography, contrast ventriculography, or radionuclide ventriculography.
* End stage renal disease requiring chronic dialysis or creatinine clearance < 20 cc/min.
* Ongoing sepsis, including active endocarditis.
* Any percutaneous coronary or peripheral interventional procedure with a bare metal or drug eluting stent performed within 30 days prior to the study procedure.
* Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 10 weeks of Heart Team assessment.
* Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
* Recent (within 6 months of Heart Team assessment) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
* Gastrointestinal (GI) bleeding that would preclude anticoagulation.
* Subject refuses a blood transfusion.
* Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
* Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbid conditions.
* Other medical, social, or psychological conditions that in the opinion of the investigator precludes the subject from appropriate consent or adherence to the protocol required follow-ups exams.
* Currently participating in an investigational drug or another device study (excluding registries).
* Evidence of an acute myocardial infarction ≤ 30 days before the study procedure.
* Need for emergency surgery for any reason.
* Liver failure (Child-Pugh class C).
* Subject is pregnant or breast feeding.

Anatomical exclusion criteria:

* Pre-existing prosthetic heart valve in any position.
* Mixed aortic valve disease (aortic stenosis with severe aortic regurgitation).
* Severe mitral regurgitation.
* Severe tricuspid regurgitation.
* Moderate or severe mitral stenosis.
* Hypertrophic obstructive cardiomyopathy.
* Echocardiographic or Multi-Slice Computed Tomography (MSCT) evidence of intracardiac mass, thrombus, or vegetation.
* Congenital bicuspid or unicuspid valve verified by echocardiography.

For transfemoral or transaxillary (subclavian) acess:

- Access vessel diameter <5.0mm or <6.0mm for patent LIMA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew R Williams, MD, Principal Investigator — New York Langone Medical Center
Locations (23):
- United States (23):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center/Medstar, Washington D.C., District of Columbia
  - St. Vincent Heart Center of Indiana/The Care Group, LLC, Indianapolis, Indiana
  - University of Kansas, Kansas City, Kansas
  - The Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconcess Medical Center, Boston, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Detroit Medical Center Cardiovascular Institute, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Morristown Memorial Hospital, Morristown, New Jersey
  - New York Langone Medical Center, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Riverside Methodist Hospital/Ohio Health Research Institute, Columbus, Ohio
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - The Methodist DeBakey Heart & Vasc Ctr/The Methodist Hosp, Houston, Texas
  - Aurora Health Care/St Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Popma JJ, Reardon MJ, Khabbaz K, Harrison JK, Hughes GC, Kodali S, George I, Deeb GM, Chetcuti S, Kipperman R, Brown J, Qiao H, Slater J, Williams MR. Early Clinical Outcomes After Transcatheter Aortic Valve Replacement Using a Novel Self-Expanding Bioprosthesis in Patients With Severe Aortic Stenosis Who Are Suboptimal for Surgery: Results of the Evolut R U.S. Study. JACC Cardiovasc Interv. 2017 Feb 13;10(3):268-275. doi: 10.1016/j.jcin.2016.08.050. PMID 28183466

RESULTS

PARTICIPANT FLOW:
Groups:
- CoreValve Evolut R TAVR System: The CoreValve Evolut R System is a transcatheter aortic valve implantation system comprised of the following three components:
  1. Evolut R Transcatheter Aortic Valve (TAV)
     >
  2. EnVeo R Delivery Catheter System (DCS) with EnVeo R InLine Sheath
     >
  3. EnVeo R Loading System (LS)
     >
     > CoreValve Evolut R TAVR system
Period: Implant
Arm/Group | CoreValve Evolut R TAVR System
Started | 241 (241 Attempted Implant)
Completed | 241 (237 Implanted)
Not Completed | 0
Period: 1-Month
Arm/Group | CoreValve Evolut R TAVR System
Started | 241 (241 Attempted Implant)
Completed | 232
Not Completed | 9
Not completed — Death | 6
Not completed — Withdrawal by Subject | 2
Not completed — Subject anesthetized but product not onsite, for medical justification treated w/commercial device | 1
Period: 6-Month
Arm/Group | CoreValve Evolut R TAVR System
Started | 232
Completed | 222
Not Completed | 10
Not completed — Death | 8
Not completed — Withdrawal by Subject | 2
Period: 12-Month
Arm/Group | CoreValve Evolut R TAVR System
Started | 213
Completed | 197
Not Completed | 16
Not completed — Death | 14
Not completed — Withdrawal by Subject | 2
Period: 24-Month
Arm/Group | CoreValve Evolut R TAVR System
Started | 197
Completed | 171
Not Completed | 26
Not completed — Death | 23
Not completed — Withdrawal by Subject | 3
Period: 36-Month
Arm/Group | CoreValve Evolut R TAVR System
Started | 171
Completed | 144
Not Completed | 27
Not completed — Death | 23
Not completed — Withdrawal by Subject | 4
Period: 48-Month
Arm/Group | CoreValve Evolut R TAVR System
Started | 144
Completed | 113
Not Completed | 31
Not completed — Death | 25
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 4
Period: 60-Month
Arm/Group | CoreValve Evolut R TAVR System
Started | 113
Completed | 109
Not Completed | 4
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — pt 103 years old no longer traveling for MD visits | 1
Not completed — Covid-19 pt not willing to be seen | 1

BASELINE CHARACTERISTICS:
Population: 241 attempted implant
Groups:
- CoreValve Evolut R TAVR System: The CoreValve Evolut R System is a transcatheter aortic valve implantation system comprised of the following three components:>
  1. Evolut R Transcatheter Aortic Valve (TAV)>
  2. EnVeo R Delivery Catheter System (DCS) with EnVeo R InLine Sheath>
  3. EnVeo R Loading System (LS)> > CoreValve Evolut R TAVR system
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165
  Male | 76
Region of Enrollment [Number; unit: participants]
  United States | 241

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality at 30 Days by Percent
Description: Percentage of patients that died by any cause at 30 days
Time Frame: Assessed at 30 days post-implantation
Population: All subjects who are brought into the procedure room and any of the following have occurred: anesthesia administered, vascular line placed, TEE placed, or any monitoring line placed.
Measure: Number (95% Confidence Interval); unit: percentage of partcipants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 241
percentage of partcipants | 2.5 [1.1 to 5.5]

2. Primary Outcome: Percentage of Patients With Disabling Stroke at 30 Days
Description: Stroke Diagnostic Criteria:
  >
  Acute episode of focal or global neurological deficit with at least 2 of the following:
  * change in level of consciousness >
  * hemiplegia, hemiparesis
  * numbness or sensory loss affecting 1 side >
  * dysphasia or aphasia
  * hemianopia
  * amaurosis fugax >
  * other neurological signs or symptoms consistent with stroke
    2.) No other readily identifiable non-stroke cause or the clinical presentation, to be determined by or in conjunctions with the designated neurologist
    3.) Confirmation of the diagnosis by at least 1 of the following:
  * Neurological specialist >
  * Neuroimaging procedure, or on clincial grounds alone > Stroke: durations of neural deficit > 24 h if available neuroimaging documents a new hemofrrhage or infarct; or the neurological deficit results in death
  Defined by VARC II:
  > An mRS (Modified Rankin Score) of 2 or more at 90 days and an increase in at least 1 mRS category from pre-stroke baseline
Time Frame: Assessed at 30 days post-implantation
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 241
percentage of participants | 3.3 [1.7 to 6.6]

3. Primary Outcome: Percent Device Success Rate Between 24 and 7 Day
Description: Percentage of patients with Device Success defined as:
  * Absence of procedural mortality, AND
  * Correct positioning of a single Evolut R valve into the proper anatomical location, AND
  * Absence of patient-prosthesis mismatch, and mean gradient , 20 mm Hg (or peak velocity < 3m/sec, AND
  * Absence of moderate or severe prosthetic valve regurgitation
Time Frame: Assessed at 24 hours to seven days post implantation
Population: All subjects implanted with the Evolut R TAV, defined as the Evolut R TAV is placed in the aortic annulus and completely released from the Enveo catheter delivery system
Measure: Number (95% Confidence Interval); unit: percentage of overall device success
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 237
percentage of overall device success | 69.2 [62.3 to 75.5]

4. Primary Outcome: Percentage of Patients With Less Than Moderate Prosthetic Regurgitation at Early Post Procedure Echocardiogram (24 Hours to 7 Days)
Description: Percentage of patience with none, trace or mild total prosthetic regurgitation at early post procedure echo cardiogram (24 hours to 7 days) as evaluated by echo core lab.
Time Frame: Assessed at 24 hours to 7 days post implantation
Population: Subset includes all subjects who are implanted with the Evolut R TAV, defined as the Evolut R TAV is placed in the aortic annulus and completely released from the Enveo catheter delivery system
Measure: Number (95% Confidence Interval); unit: percentage of partcipants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 237
percentage of partcipants | 96.5 [93.3 to 98.5]

5. Secondary Outcome: Individual Component of VARC II Safety Endpoint: Percentage of People Requiring Valve-related Dysfunction Requiring Repeat Procedure (BAV, TAVI, or SAVR)
Description: Percentage of patients with any valve dysfunction that requires repeat procedure (e.g. balloon valvuloplasty, TAVI, or surgical AVR), per VARC II definition.
Time Frame: Assessed at 30 days post-implantation
Population: The safety subset includes all subjects who are brought into the procedure room and any of the following have occurred: anesthesia administered, vascular line placed, or any monitoring line placed.
Measure: Number (95% Confidence Interval); unit: percentage of overall patients
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 241
percentage of overall patients | 0.0 [0.0 to 1.6]

6. Secondary Outcome: Coronary Artery Obstruction Requiring Intervention.
Description: Angiographic or echocardiographic evidence of a new, partial or complete, obstruction of a coronary ostium, either by the Evolut R prosthesis itself, the native leaflets, calcifications, or dissection, occurring during or after the TAVI procedure.
Time Frame: Assessed at 30 days post-implantation
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 241
percentage of participants | 0.4 [0.1 to 3.0]

7. Secondary Outcome: Percent VARC II Combined Safety Endpoint at 30 Days
Description: VARC II composite safety endpoint rate includes percent freedom from the following components:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury: stage 2 or 3 (including renal replacement therapy).
  * Coronary artery obstruction requiring intervention.
  * Major vascular complication.
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR)
Time Frame: Assessed at 30 days post-implantation
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 241
percentage of participants | 14.5 [10.6 to 19.7]

8. Secondary Outcome: Percent of Patients With Acute Kidney Injury: Stage 2 or 3 (Including Renal Replacement Therapy).
Description: Stage 2
  1. Increase in serum creatinine to 200%-299% (2.0%-2.99% increase compared with baseline) OR
     >
  2. Urine output <0.5 mL/kg/h for >12 but <24 h > Stage 3 >
  1) Increase in serum creatinine to ≥300% (>3 x increase compared with baseline) OR serum creatinine of ≥4.0 mg/dL (≥354 mmol/L) with an acute increase of at least 0.5 mg/dL (44 mmol/L) OR
  * Urine output <0.3 ml/kg/h for ≥24 h OR
    >
  * Anuria for ≥12 h
Time Frame: Assessed at 30 days post-implantation
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 241
percentage of participants | 1.3 [0.4 to 3.9]

9. Secondary Outcome: Percentage of Patients With Life-threatening or Disabling Bleeding Event Rate
Description: 1. Fatal bleeding (BARC type 5) OR
     >
  2. Bleeding in a critical organs, such as intracranial, intraspinal,
     > intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome (BARC type 3b and 3c) OR
     >
  3. Bleeding causing hypovolemic shock or severe hypotension requiring vasopressors or surgery (BARC type 3b) OR
     >
  4. Overt source of bleeding with drop in hemoglobin ≥5 g/dL or whole blood or packed red blood cells (RBCs) transfusion ≥4 units* > (BARC type 3b)
Time Frame: Assessed at 30 days post-implantation
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 241
percentage of participants | 7.1 [4.4 to 11.2]

10. Secondary Outcome: Percent Rate of Patients Who Received New Permanent Pacemaker Implant at 30 Days
Description: Percent of patients who underwent implantation of new permanent pacemaker or ICD during or after index procedure
Time Frame: Assessed at 30 days
Population: All subjects who are brought into the procedure room and any of the following have occurred: anesthesia administered, vascular line placed, TEE placed, or any monitoring line placed. Additionally, these patients did NOT have ICD or PPM at the time of the index procedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 201
percentage of participants | 19.7 [14.7 to 26.1]

11. Secondary Outcome: Percent Resheath and Recapture Success Rate
Description: Resheath or recapture success rate (where attempted) where a successful resheath is defined as the intended portion of the Evolut R is resheathed into the capsule of the delivery catheter to the intended amount, as verified by flouroscopy; and a successful recapture is defined as the entire Evolut R TAV (including the frame) is full resheathed into the capsule of the delivery catheter until there is no gap between the capsule and the tip , as verified by flouroscopy. Resheath or recapture wa attempted in a subset of patients. Success rate is calculated as successful resheath or recaputure events in the number of total events. Resheath anad recapture is only possible during the index procedure.
Time Frame: Assessed intra-procedurally
Population: 65 patients had resheath or recapture feature used during the 241 attempted procedures.
Measure: Number; unit: percentage of resheath or recapture
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 65
percentage of resheath or recapture | 96.9

12. Secondary Outcome: Hemodynamic Performance -Mean Gradient
Description: Mean gradient by Doppler echocardiography.
Time Frame: Assessed at baseline, 30 days, 6 months, and 1 year
Population: The Implanted population consisted of all As Treated Subjects who underwent an index procedure and were implanted with the Evolut R system. Only subjects with echo can be analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 237
mmHg
  baseline | 48.2 (13.0)
  30 days: number analyzed (Participants) | 228
  30 days | 7.8 (3.1)
  6 months: number analyzed (Participants) | 208
  6 months | 8.4 (3.8)
  1 year: number analyzed (Participants) | 191
  1 year | 9.1 (4.7)

13. Secondary Outcome: Major Vascular Complication
Description: 1. Any aortic dissection, aortic rupture, annulus rupture, left ventricle perforation, or new apical aneurysm/pseudoaneurysm OR
     >
  2. Access-related vascular injury (dissection, stenosis, perforation, rupture, arterio-venous fistula, pseudoaneurysm, hematoma, irreversible nerve injury, compartment syndrome, percutaneous closure device failure) leading to death, life-threatening or major bleeding, visceral ischemia, or neurological impairment OR
     >
  3. Distal embolization (noncerebral) from a vascular source requiring surgery or resulting in amputation or irreversible end-organ damage OR
     >
  4. The use of unplanned endovascular or surgery associated with death, major bleeding, visceral ischemia or neurological impairment OR
     >
  5. Any new ipsilateral lower extremity ischemia documented by patient symptoms, physical exam, and/or decreased or absent blood flow on lower extremity angiogram OR
     >
  6. Surgery for access site nerve injury OR
     >
  7. Permanent access related nerve injury
Time Frame: Assessed at 30 days post-implantation
Population: The Implanted population consisted of all As Treated Subjects who underwent an index procedure and were implanted with the Evolut R system.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 237
percentage of participants | 7.5 [4.8 to 11.7]

14. Secondary Outcome: Hemodynamic Performance - Aortic Valve Area
Description: Hemodynamic performance by Doppler echocardiography - Aortic Valve Area cm2
Time Frame: Assessed at baseline, 30 days, 6 months, and 1 year
Population: The hemodynamic performance subset includes all subjects implanted with the Evolut R TAV for more than 24 hours post implantation - only subjects with echo can be analyzed.
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 237
cm²
  baseline: number analyzed (Participants) | 211
  baseline | 0.6 (0.2)
  30 days: number analyzed (Participants) | 204
  30 days | 1.9 (0.5)
  6 months: number analyzed (Participants) | 180
  6 months | 1.8 (0.5)
  1 year: number analyzed (Participants) | 160
  1 year | 1.8 (0.5)

15. Secondary Outcome: Hemodynamic Performance: Total Prosthetic Valve Regurgitation Graded as Moderate or Severe
Description: Hemodynamic performance: the percent of patients who have a degree of total prosthetic valve regurgitation that is moderate or severe.
Time Frame: Assessed at 30 days, 6 months, and 1 year
Population: The hemodynamic performance subset includes all subjects implanted with the Evolut R TAV for more than 24 hours post implantation. Only subjects with echo can be analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | CoreValve Evolut R TAVR System
Number analyzed (Participants) | 237
percentage of participants
  30 days: number analyzed (Participants) | 227
  30 days | 5.7
  6 months: number analyzed (Participants) | 205
  6 months | 5.4
  1 year: number analyzed (Participants) | 191
  1 year | 3.7

ADVERSE EVENTS:
Time Frame: All events - 12 months, All Cause Mortality - 60 months
Groups:
- CoreValve Evolut R TAVR System: The CoreValve Evolut R System is a transcatheter aortic valve implantation system comprised of the following three components:
  Evolut R Transcatheter Aortic Valve (TAV) EnVeo R Delivery Catheter System (DCS) with EnVeo R InLine Sheath EnVeo R Loading System (LS)
Arm/Group | CoreValve Evolut R TAVR System
All-Cause Mortality (participants affected / at risk) | 107/241
Serious Adverse Events (participants affected / at risk) | 170/241
Other Adverse Events (participants affected / at risk) | 197/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoreValve Evolut R TAVR System (N=241)
Anaemia (Blood and lymphatic system disorders) | 36 (39)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1)
Splenic Infarction (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3)
Angina Unstable (Cardiac disorders) | 1 (1)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 15 (16)
Atrioventricular Block Complete (Cardiac disorders) | 32 (32)
Atrioventricular Block Second Degree (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 2 (2)
Bundle Branch Block Left (Cardiac disorders) | 4 (4)
Bundle Branch Block Right (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 4 (4)
Cardiac Failure (Cardiac disorders) | 6 (6)
Cardiac Failure Acute (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 22 (28)
Cardiac Perforation (Cardiac disorders) | 3 (3)
Cardiogenic Shock (Cardiac disorders) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 4 (4)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1)
Nodal Rhythm (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1)
Right Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Right Ventricular Failure (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 3 (3)
Sinus Node Dysfunction (Cardiac disorders) | 2 (2)
Stress Cardiomyopathy (Cardiac disorders) | 1 (1)
Ventricular Asystole (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Cataract (Eye disorders) | 2 (2)
Glaucoma (Eye disorders) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 2 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 12 (12)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 4 (4)
Intestinal Ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 4 (5)
Chest Pain (General disorders) | 3 (3)
Death (General disorders) | 2 (2)
Device Deployment Issue (General disorders) | 1 (1)
Device Dislocation (General disorders) | 1 (1)
Implant Site Haemorrhage (General disorders) | 3 (4)
Implant Site Pain (General disorders) | 1 (1)
Lead Dislodgement (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Gallbladder Disorder (Hepatobiliary disorders) | 1 (1)
Abdominal Wall Abscess (Infections and infestations) | 1 (1)
Acquired Immunodeficiency Syndrome (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 5 (5)
Diverticulitis (Infections and infestations) | 1 (1)
Diverticulitis Intestinal Haemorrhagic (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Incision Site Infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 12 (16)
Pneumonia Staphylococcal (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 8 (8)
Septic Shock (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 9 (9)
Urosepsis (Infections and infestations) | 1 (2)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Arterial Injury (Injury, poisoning and procedural complications) | 2 (2)
Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Feeding Tube Complication (Injury, poisoning and procedural complications) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 3 (3)
Incision Site Complication (Injury, poisoning and procedural complications) | 4 (4)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 6 (7)
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Blood Magnesium Decreased (Investigations) | 2 (2)
Blood Pressure Increased (Investigations) | 1 (1)
International Normalised Ratio Increased (Investigations) | 2 (2)
Urine Output Decreased (Investigations) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small Intestine Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Brain Injury (Nervous system disorders) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 10 (12)
Dizziness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Hemiplegia (Nervous system disorders) | 1 (1)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 3 (3)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1)
Speech Disorder (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Thalamic Infarction (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 4 (5)
Delirium (Psychiatric disorders) | 1 (1)
Hallucination, Visual (Psychiatric disorders) | 1 (1)
Mental Disorder (Psychiatric disorders) | 4 (4)
Acute Kidney Injury (Renal and urinary disorders) | 5 (6)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Renal Infarct (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 2 (3)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Subacute Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (18)
Aortic Dissection (Vascular disorders) | 1 (1)
Aortic Dissection Rupture (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Femoral Artery Dissection (Vascular disorders) | 2 (2)
Femoral Artery Occlusion (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 9 (9)
Hypotension (Vascular disorders) | 16 (16)
Iliac Vein Occlusion (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 1 (1)
Labile Blood Pressure (Vascular disorders) | 3 (3)
Labile Hypertension (Vascular disorders) | 1 (1)
Malignant Hypertension (Vascular disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (2)
Peripheral Artery Dissection (Vascular disorders) | 1 (1)
Peripheral Artery Stenosis (Vascular disorders) | 2 (2)
Peripheral Ischaemia (Vascular disorders) | 3 (3)
Peripheral Vascular Disorder (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoreValve Evolut R TAVR System (N=241)
Anaemia (Blood and lymphatic system disorders) | 48 (49)
Leukocytosis (Blood and lymphatic system disorders) | 19 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 37 (37)
Atrial Fibrillation (Cardiac disorders) | 19 (21)
Atrioventricular Block First Degree (Cardiac disorders) | 39 (40)
Bundle Branch Block Left (Cardiac disorders) | 79 (82)
Bundle Branch Block Right (Cardiac disorders) | 13 (13)
Cardiac Failure Congestive (Cardiac disorders) | 16 (17)
Ventricular Extrasystoles (Cardiac disorders) | 13 (13)
Chest Pain (General disorders) | 13 (14)
Urinary Tract Infection (Infections and infestations) | 32 (38)
Fall (Injury, poisoning and procedural complications) | 18 (25)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 16 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (16)
Acute Kidney Injury (Renal and urinary disorders) | 17 (17)
Renal Failure (Renal and urinary disorders) | 13 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 27 (29)
Hypertension (Vascular disorders) | 40 (44)
Hypotension (Vascular disorders) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No